CLINICAL TRIAL: NCT01949220
Title: International Post-Marketing Surveillance of Willfact-Wilfactin in Patients With Inherited Von Willebrand Disease.
Brief Title: Willebrand International Non-interventional Global Surveillance
Status: Completed | Type: Observational
Sponsor: Laboratoire français de Fractionnement et de Biotechnologies (Industry)
Responsible Party: Sponsor
Other Study IDs: WINGS
Record Dates: First submitted 2013-09-10; First posted 2013-09-24 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2017-12

CONDITIONS: Von Willebrand Disease
Keywords: Inherited; Von Willebrand disease; Von Willebrand factor; Deficiency; safety
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Von Willebrand factor deficient patient: Inherited von Willebrand disease

SUMMARY:
Collect information about WILLFACT or WILFACTIN in their real life clinical use and identify the therapeutic practices in an international environment.

DETAILED DESCRIPTION:
Non-interventional, prospective, non comparative, international, multicentre study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inherited von Willebrand disease
* Patients treated with WILLFACT or WILFACTIN
* Patient or parent/legal representative who has provided written signed and dated informed consent before any data collection.

Exclusion Criteria:

* Patients who usually do not keep injection log up to date, when treated.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient, whatever their age, with inherited von Willebrand disease
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Documentation of product consumption data | at each follow-up visit, up to 24 months
  Product consumption (VWF International Units) by analysis of posology, frequency in relation to the severity of bleeding, type of surgery and other clinical situations.

SECONDARY OUTCOMES:
Collection and analysis of adverse events and VWF immunological safety | at each follow-up visit, up to 24 months
  Adverse event (type, seriousness, severity, frequency, outcome), anti VWF-antibody and anti FVIII-antibody.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang MIESBACH, Dr, Study Director — Medizinische Klinik III, Goethe Universitat, D-60590 Frankfurt/Main (Germany); Flora PEYVANDI, Prof., Study Director — Faculty of Medicine, University of Milan, 20122 Milan (Italy)
Locations (18):
- Belgium (2):
  - Hopital des enfants Reine Fabiola, Antwerp
  - UZA hopital universitaire, Edegem
- University Hospital, Brno, Czechia
- University Central Hospital, Helsinki, Finland
- Germany (9):
  - Charité Universitätsmedizin, Berlin
  - GZRR Gerinnungszentrum Rhein/ Ruhr, Duisburg
  - Universitatsklinikum, Essen
  - Goethe Universitat, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
  - Werlhof-Institut für Hämostaseologie GmbH, Hanover
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Universitatsklinikum, Mainz
  - Klinikum der Universität, München
- Hemophilia center "LAIKO" general hospital, Athens, Greece
- Italy (3):
  - Centro di Riferimento Regionale per Emofilia e Trombosi, Catania
  - AOUC- Azienda Ospedaliero-Universitaria Carregi, Florence
  - University of Milan, Milan
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No